CLINICAL TRIAL: NCT00463125
Title: Platelet Gel for Digital Ulcers in Patients With SSc: a Randomized Controlled Trial
Brief Title: Platelet Gel in Systemic Sclerosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università Politecnica delle Marche (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UPM13746IC
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Scleroderma, Systemic
Keywords: Scleroderma, systemic; therapeutic; platelet gel
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Platelet Gel

SUMMARY:
* Systemic sclerosis (scleroderma; SSc) is a connective tissue disease characterized by a progressive fibrosis of the skin and visceral organs.
* A diffuse cutaneous microvascular damage occurs in 30-50% of patients, often leading to digital ulcers development, responsible for pain, functional disability, disfiguring scars, digital bony reabsorption, infection and osteomyelitis.
* Although the availability of drugs as i.v. prostacyclin analogs, oral vasodilating agents, oral phosphodiesterase-5 inhibitors, oral endothelin receptor blockers has improved the prognosis, digital ulcers are frequently refractory to the medical treatment.
* Preliminary data seems to demonstrate a pivotal role played by some growth factors (PDGF, TGF beta 1-2, IGF) in the process of ulcers healing: tissue regeneration and re-epithelization. Alpha-granules in the platelets store these factors in significant amount.
* Recently, the application of a gel rich in platelets, prepared from donors' plasma taken by apheresis, seems to be beneficial to enhance pressure and vascular ulcers healing.
* On the basis of these considerations we expect that application of a platelet gel, combined with advanced dressing and conventional medical therapy, makes a more rapid healing of digital ulcers in patients with systemic sclerosis. We decided to conduct a double blind RCT to test this hypothesis

ELIGIBILITY:
Inclusion Criteria:

* Digital ulcers (NPUAP stage≥2) in patients with SSc (ACR criteria)
* Current medical treatment with intravenous prostanoids
* Availability to come to our centre for weekly ulcer assessment and medication
* Capacity to give informed consent

Exclusion Criteria:

* Clinical evidence of skin infection
* Current treatment with Bosentan or Sildenafil
* Presence of necrotic material occluding the wound bed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2007-03; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Time from diagnosis to complete ulcer healing
Rate of ulcers healed during the follow up period (10 weeks)

SECONDARY OUTCOMES:
Rate of ulcers healed during the follow up period (10 weeks)
Pain evaluation (VAS scale)
Rate of complications

CONTACTS AND LOCATIONS:
Overall Officials: Armando Gabrielli, MD, professor, Study Director — Università Politecnica delle Marche
Locations (1):
- Università politecnica delle marche, Ancona, Italy